CLINICAL TRIAL: NCT05584527
Title: Assessment of the Effects of a 24-hour Cold and Heat Exposure on the Factors Influencing Food Intake
Acronym: TEMPCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PBMD08; 2022-A01862-41 (Other: IDRCB)
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Eating Habit; Cold Exposure; Heat
Keywords: Heat Exposure; Food Intake
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva and blood samples will be collected during each experimental visit :
  * saliva samples will be collected to measure salivary cortisol level.
  * blood samples will be collected to measure plasma levels of acylated ghrelin, leptin, peptide YY and Glucagon-like peptide-1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Heat exposure (32°C) — The participants will be exposed to heat (32°C) for 24 hours in a climatic apartment.
  During the exposure,
  * food intake and energy expenditure will be measured
  * several physiological tests will be performed: hunger and thirst questionnaires, thermal sensations, skin temperature measurement, weighing, olfactory and gustatory capacities, food preference questionnaire, etc.
  * sleep brain activity will be monitored using a headband
  * urine and saliva samples will be collected.
Other: Cold exposure (16°C) — The participants will be exposed to cold (16°C) for 24 hours in a climatic apartment.
  During the exposure,
  * food intake and energy expenditure will be measured
  * several physiological tests will be performed: hunger and thirst questionnaires, thermal sensations, skin temperature measurement, weighing, olfactory and gustatory capacities, food preference questionnaire, etc.
  * sleep brain activity will be monitored using a headband
  * urine and saliva samples will be collected.
Other: Thermoneutral exposure (24°C) — The participants will be exposed to a thermoneutral environment (24°C) for 24 hours in a climatic apartment.
  During the exposure,
  * food intake and energy expenditure will be measured
  * several physiological tests will be performed: hunger and thirst questionnaires, thermal sensations, skin temperature measurement, weighing, olfactory and gustatory capacities, food preference questionnaire, etc.
  * sleep brain activity will be monitored using a headband
  * urine and saliva samples will be collected.

SUMMARY:
Military personnel and athletes have a very high energy expenditure which is increased during certain key periods (intense training, competition and mission). Compensating for this expenditure through food can be complicated by physiological ingestive limits and logistical and organizational constraints (number of meals, availability of food), which leads these populations to regularly experience energy deficit situations (intake below requirements), which could alter physical and cognitive performance and major physiological functions.

Among the many constraints to which military personnel and athletes are exposed to (stress, sleep deprivation, travel, etc.) that can increase the risk of energy deficits, the impact of thermal environmental constraints is not well known. The seasonal impact and travel to countries with very different thermal environments can lead these populations to experience cold and hot conditions for long periods.

Understanding how heat and cold exposure modifies appetite and energy intake therefore appears to be of great importance.

The hypothesis of this study is that a 24 h heat exposure would produce a rapid and long-lasting anorexigenic action impacting energy intake, while a cold exposure would produce the opposite effect (orexigenic action).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18 to 40 years old
* Active (≥ 3 hours of physical activity per week)
* Healthy (no metabolic pathology)
* Affiliated to the social security system
* Having given written consent to participate.

Exclusion Criteria:

* Unusual eating pattern (< 3 meals per day) or irregular eating pattern
* Pattern of dietary restriction (determined by the Three-Factor Eating Questionnaire-21)
* Unusual sleep pattern (Epworth score > 10, insomnia severity score > 14, Pittsburgh Sleep Quality Index > 5), sleep duration < 6 h per night or difficulty falling asleep)
* Metabolic pathology
* On medication
* Previously exposed to unusual levels of heat or cold (vacation, missions) in the 4 months prior to inclusion
* Refusal to participate.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be composed of young and healthy men.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Total energy intake (in kilojoules) measured at the end of each condition (heat exposure, cold exposure and thermoneutral exposure) | Through study completion (30 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided